CLINICAL TRIAL: NCT05390619
Title: Comparison of Different Doses of Verteporfin Photodynamic Therapy in the Treatment of Chronic Central Serous Chorioretinopathy
Brief Title: Different Doses of vPDT in the Treatment of cCSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yao Yiou, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDL2020-04
Record Dates: First submitted 2022-05-17; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Central Serous Chorioretinopathy; Therapy, Photodynamic
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50% dose of PDT (Experimental): Patients received 50% dose of verteporfin PDT therapy.
  Interventions: Procedure: 50% dose of photodynamic therapy
- 70% dose of PDT (Experimental): Patients received 70% dose of verteporfin PDT therapy.
  Interventions: Procedure: 70% dose of photodynamic therapy

INTERVENTIONS:
Procedure: 50% dose of photodynamic therapy — Verteporfin (Visudyne; Novartis, Switzerland) was administrated intravenously over 10 minutes with 50% doses based on the randomization . Fifteen minutes after commencing the verteporfin infusion, a contact lens (Volk® area centralis) was positioned on the affected eye, the treatment area was exposed to a 689 nm laser with a fluence of 600 mw/cm2 for 83 seconds and a total laser energy of 50 J/cm2.
  Arms: 50% dose of PDT
Procedure: 70% dose of photodynamic therapy — Verteporfin (Visudyne; Novartis, Switzerland) was administrated intravenously over 10 minutes with 70% doses based on the randomization . Fifteen minutes after commencing the verteporfin infusion, a contact lens (Volk® area centralis) was positioned on the affected eye, the treatment area was exposed to a 689 nm laser with a fluence of 600 mw/cm2 for 83 seconds and a total laser energy of 50 J/cm2.
  Arms: 70% dose of PDT

SUMMARY:
This is a prospective, randomized and controlled clinical trial of photodynamic therapy (PDT) for chronic central serous chorioretinopathy (CSC). The patients who met the inclusion criteria were randomly divided into 50% dose PDT treatment group and 70% dose PDT treatment group. The primary treatment success rate and adverse event rate of the two groups were compared by optical coherence tomography (OCT), and then the best PDT treatment scheme for chronic CSC was summarized.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, regardless of gender;
* Meet the diagnostic criteria of central serous chorioretinopathy;
* The course of CSC (subject to the symptoms of this disease) is more than 3 months;
* Patients with simultaneous diseases of both eyes were included in those with more subretinal fluid.

Exclusion Criteria:

* macular neuroretinal detachment caused by rhegmatogenous retinal detachment, uveitis, age-related macular degeneration, polypoid choroidal angiopathy and other fundus diseases;
* a previous history of PDT treatment;
* systemic hormone or local hormone nasal spray is being used, or hormone is stopped for less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The complete absorption rate of subretinal fluid | 3 months after the primary PDT
  The absorption of subretinal fluid was observed on optical coherence tomography at each follow up visit

SECONDARY OUTCOMES:
Central foveal thickness change after the PDT | 12 months after the PDT
  The hight of central foveal thickness was measured on optical coherence tomography at each visit
Subfoveal choroidal thickness change after the PDT | 12 months after the PDT
  The hight of Subfoveal choroidal thickness was measured on optical coherence tomography at each visit
Best corrected visual acuity change after the PDT | 12 months after the PDT
  The BCVA was tested at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Yuou Yao, Dr, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China